CLINICAL TRIAL: NCT02529475
Title: Evaluation of Inner Ear and Brain Structures With Contrast-enhanced MRI in Healthy Subjects (HYDROPS)
Acronym: HYDROPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment problem-covid-
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.428
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Meniere Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gadoteric acid (Experimental): Gadoteric acid 0.2 mmol/kg
  Interventions: Drug: Gadoteric acid

INTERVENTIONS:
Drug: Gadoteric acid — Comparison with patients with Meniere's disease

SUMMARY:
* This prospective study aims to better characterize inner ear's perilymphatic structures with Magnetic Resonance Imaging using contrast media and delayed injection in healthy subjects
* MR Perfusion Imaging will be assess in both cochlea as well
* Primary auditory brain pathways will be evaluated through MR diffusion imaging

ELIGIBILITY:
Inclusion Criteria:

* Major subjects of over 40 years (mean age of Meniere's disease 40 to 50 years)
* Informed consent signed
* Medical examination performed prior to participation in research
* Patients without history of inner ear disease
* Recipient of a French social security scheme

Exclusion Criteria:

* Patients minors
* Patients on a legal protection regime type guardianship
* Respiratory pathologies, cardiovascular, renal, diabetes
* Claustrophobia
* Contraindications to exposure to a magnetic field
* Contraindications to injecting Dotarem ®

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Gadolinium enhancement in inner ear structures as measured by MR T1 Weighted Imaging | One MR scan (4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud ATTYE, PH, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - GrenobleUniversityHospital, Grenoble
  - Hôpital Lariboisière, Paris
  - Hôpital Charles Nicolle, Rouen

REFERENCES:
- [Derived] Eliezer M, Maquet C, Horion J, Gillibert A, Toupet M, Bolognini B, Magne N, Kahn L, Hautefort C, Attye A. Detection of intralabyrinthine abnormalities using post-contrast delayed 3D-FLAIR MRI sequences in patients with acute vestibular syndrome. Eur Radiol. 2019 Jun;29(6):2760-2769. doi: 10.1007/s00330-018-5825-0. Epub 2018 Nov 9. PMID 30413960